CLINICAL TRIAL: NCT06716658
Title: Exploratory Clinical Study of JAK1 Inhibitor Golidocitnib in the Treatment of Relapsed/Refractory Indolent T/NK-Cell Lymphomas：An Open, Prospective, Exploratory Clinical Trial
Brief Title: JAK1 Inhibitor Golidocitnib for the Treatment of Relapsed/Refractory Indolent T/NK-cell Lymphomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Tianjin First Central Hospital (Other); The First Affiliated Hospital of Air Force Medicial University (Other); The First Hospital of Jilin University (Other); The First Affiliated Hospital of Nanchang University (Other); Henan Cancer Hospital (Other Government); Second Xiangya Hospital of Central South University (Other); Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024084
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Lymphoma, T-Cell; NK-LGL Leukemia; T-LGL Leukemia; Cutaneous T Cell Lymphoma; Cutaneous T Cell Lymphoma (CTCL); Large Granular Lymphocyte Leukemia; Large Granular Lymphocytic Leukemia; Indolent T-Cell Lymphoproliferative Disorder of the Gastrointestinal Tract; Primary Cutaneous Acral CD8-Positive T-Cell Lymphoma; Mycosis Fungoides
Keywords: Indolent T/NK-cell lymphomas; JAK1 inhibitor
MeSH Terms: conditions — Lymphoma, T-Cell; Leukemia, Large Granular Lymphocytic; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JAK1 inhibitor (Experimental): Golidocitnib 150mg QD orally
  Interventions: Drug: JAK1 Inhibitor

INTERVENTIONS:
Drug: JAK1 Inhibitor — Golidocitnib 150mg QD orally, with a 28-day cycle. Efficacy will be evaluated once per cycle during the first year, and once every two cycles thereafter. Treatment will continue for up to 24 cycles, or until disease progression, lack of response within the first 6 cycles, or the occurrence of intolerable toxicity, whichever occurs first

SUMMARY:
Indolent T/NK-cell lymphomas are a heterogeneous group of lymphoproliferative diseases originating from T/NK cells, characterized by slow growth and proliferation, but currently remain incurable. For indolent T/NK-cell lymphomas that are unresponsive to first-line treatment, there are few treatment options available and the prognosis is poor. This study is an open-label, prospective clinical trial aimed at evaluating the feasibility, efficacy, and safety of PI3K inhibitors in the treatment of relapsed/refractory indolent T/NK-cell lymphomas. Patients will be treated with Golidocitnib, with an expected overall response rate of 60% for JAK1 inhibitor Golidocitnib treatment.

DETAILED DESCRIPTION:
Plan to enroll 48 patients with relapsed/refractory indolent T/NK-cell lymphomas; they will receive JAK1 inhibitor treatment (Golidocitnib150mg QD orally, with a 28-day cycle). Efficacy will be evaluated once per cycle during the first year, and once every two cycles thereafter. Treatment will continue for up to 24 cycles, or until disease progression, lack of response within the first 6 cycles, or the occurrence of intolerable toxicity, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, with no restrictions on gender;
2. Histologically confirmed relapsed/refractory (R/R) indolent T/NK-cell; lymphoma that has failed at least one systemic therapy or is intolerant to such treatment and/or currently has no effective standard treatment options;
3. The patient meets the criteria for appropriate therapeutic indications;
4. ECOG performance status of 0-2;
5. Adequate organ function, defined as: Total bilirubin (TBIL) ≤ 1.5 × ULN; ALT and AST ≤ 2.5 × ULN; Blood urea nitrogen (BUN)/Urea and creatinine (Cr) ≤ 1.5 × ULN; Left ventricular ejection fraction (LVEF) ≥ 50%; Fridericia-corrected QT interval (QTcF): < 450 ms for males, < 470 ms for females;
6. An expected survival time of at least 3 months;
7. Male and female subjects of childbearing potential must agree to use effective contraception throughout the study period and for 6 months after the last dose of the investigational drug;
8. A washout period of ≥ 4 weeks since receiving any prior antitumor therapies (including radiotherapy, chemotherapy, hormone therapy, surgery, or molecular targeted therapy) before participating in this study;
9. The subject has not participated in any other clinical trial within 1 month prior to enrollment;
10. The subject agrees to and signs the informed consent form.

Exclusion Criteria:

1. Subjects who have previously used any JAK inhibitors;
2. Subjects with clinical conditions such as dysphagia, malabsorption, or other chronic gastrointestinal diseases that may interfere with compliance and/or absorption of the study drug;
3. Subjects with active viral, bacterial, or fungal infections requiring treatment (e.g., pneumonia);
4. Subjects with HBV or HCV infections, defined as HBsAg and/or HBcAb positivity and HBV DNA copy number ≥ the upper limit of normal (ULN), or acute or chronic active hepatitis C (HCV antibody-positive);
5. Subjects with a history of immunodeficiency, including those who are HIV-positive, or those with other acquired or congenital immunodeficiency diseases, a history of organ transplantation, or a history of allogeneic bone marrow or hematopoietic stem cell transplantation;
6. Subjects who have undergone autologous hematopoietic stem cell transplantation within 90 days prior to the first dose of study treatment;
7. Subjects with severe or uncontrolled cardiovascular diseases;
8. Subjects with severe concomitant diseases that pose a significant risk to patient safety or, in the investigator's judgment, may interfere with the completion of the study (e.g., uncontrolled hypertension, diabetes, or thyroid disorders);
9. Pregnant or breastfeeding female subjects, or baseline positive pregnancy test results in women of childbearing potential;
10. Subjects with a history of other malignancies diagnosed or treated within the past 5 years;
11. Any other conditions that, in the investigator's opinion, render the subject unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | up to 5 years
  complete remission rate + partial remission rate

SECONDARY OUTCOMES:
The safety of JAK1 inhibitor | up to 5 years
  Incidence of adverse events, serious adverse events and significant adverse event
Complete remession rate | up to 5 years
  Hematological PR was defined as an improvement in blood counts ANC > 0.5 × 109/L; HGB increased by >1 g/dL; PLT > 50 × 109/L
Duration of remission | up to 5 years
  the time from response to progression/death (P/D)
Time to response | up to 5 years
  from the start of treatment to the first observed partial remission
Progression-free survival | up to 5 years
  the time from treatment initiation until disease progression or death
Overall survival | up to 5 years
  The time from the start of treatment to the patient's death from any cause
Disease control rate | up to 5 years
  the proportion of patients whose tumors have not progressed after treatment over a specific period of time. Specifically, DCR includes the percentage of patients who achieve complete response (CR), partial response (PR), and stable disease (SD).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Institute of Hematology & Blood Diseases Hospital, China, Tianjin, Tianjin Municipality
  - Institute of Hematology & Blood Diseases Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No